CLINICAL TRIAL: NCT01172795
Title: Diffuse Noxious Inhibitory Controls (DNIC): Nociceptive Modulation and Interaction With Neurocognitive Performance in Chronic Pain
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Vrije Universiteit Brussel (Other)
Collaborators: Research Foundation Flanders (Other)
Other Study IDs: B-Cognitive tests
Record Dates: First submitted 2010-07-29; First posted 2010-07-30 (Estimated); Last update posted 2010-07-30 (Estimated); Status verified 2010-07

CONDITIONS: Fibromyalgia; Whiplash; Chronic Pain
Keywords: Whiplash associated disorder; chronic pain; neural inhibition; neuropsychological tests
MeSH Terms: conditions — Fibromyalgia; Whiplash Injuries; Chronic Pain

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional

GROUPS / COHORTS (3):
- healthy controls
  Interventions: Behavioral: Relaxation session; Behavioral: Neurocognitive test battery
- chronic whiplash patients
  Interventions: Behavioral: Relaxation session; Behavioral: Neurocognitive test battery
- Fibromyalgia patients
  Interventions: Behavioral: Relaxation session; Behavioral: Neurocognitive test battery

INTERVENTIONS:
Behavioral: Relaxation session — 30 minutes relaxation session (audiotape)
Behavioral: Neurocognitive test battery — the psychomotor vigilance task, span task and the stroop task on computer

SUMMARY:
Diffuse noxious inhibitory control In order to quantify central sensitization in chronic pain patients, the Diffuse Noxious Inhibitory Control (DNIC) model has been used frequently. DNIC relies on painful conditioning stimulation of one part of the body to inhibit pain in another part, to remove the "noise" and to focus on relevant stimuli.

Earlier studies provided evidence for malfunctioning of DNIC in Fibromyalgia (FM) patients. However, the cause of this impairment is not yet elucidated, and further study is required to unravel the pathophysiology of DNIC in FM.

Hypothalamus-Pituitary-Adrenal (HPA) axis Besides neural mechanisms, also hormonal abnormalities could cause altered pain processing. Cortisol is released in answer to pain to suppress the pain. Given the evidence for hypofunction of the hypothalamic-pituitary-adrenal axis and the lower cortisol release in response to stressors in a proportion of FM patients and in chronic whiplash associated disorders (WAD) patients, the relation between pain and cortisol in these patients may be an interesting topic to consider.

Neurocognitive performance Besides chronic pain, people with chronic WAD and FM suffer from severe concentration difficulties and decreased neurocognitive capabilities (reduced reaction time, short term memory deficits etc. The decreased neurocognitive performance is known to be related to pain severity in various chronic pain populations. It is hypothesized that malfunctioning of descending inhibitory pathways and subsequent chronic pain experience precludes optimal neurocognitive performance.

Objectives The present investigation addresses the (patho)physiological mechanisms of DNIC in chronic pain populations.

1. Firstly, patients with FM, chronic WAD and healthy controls are compared regarding functioning of DNIC, cortisol levels and response and neurocognitive performance (case-control).
2. Secondly, the possible interaction between the functioning of DNIC, cortisol and neurocognitive performance is studied in patients with FM, WAD and healthy control subjects (cross-sectional).
3. Thirdly, to examine whether a fatiguing neurocognitive stressor changes DNIC and cortisol levels in patients with FM, chronic WAD or healthy sedentary control subjects.

ELIGIBILITY:
Inclusion Criteria:

* 30 FM group: comply with the diagnostic criteria for FM as defined by the American College of Rheumatology.
* 30 WAD group: comply with the criteria of the Quebec Task Force (grade I to III)
* 40 healthy pain-free control subjects
* Dutch speaking
* aged between 18 and 65 years.

Exclusion Criteria:

* FM patients reporting a history of a whiplash trauma
* WAD patients fulfilling the diagnostic criteria for FM
* healthy control subjects cannot suffer any pain complaints
* cannot be pregnant or until 1 year postnatal
* asked to stop analgesics 48 hours prior to study participation, not to undertake physical exertion, and to refrain from consuming caffeine, alcohol or nicotine on the day of the experiment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Thirty patients with FM, 30 patients with WAD and 30 healthy pain-free control subjects will be enrolled. All three groups will be comparable for age, gender, education level and socioeconomic status; both patient groups will be comparable for illness duration. Sample size was calculated based on a power analysis (0.80), based on the assumption of a 20% difference of DNIC functioning after neurocognitive testing.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-07; Primary Completion 2011-07 (Estimated); Study Completion 2011-08 (Estimated)

PRIMARY OUTCOMES:
pain inhibition efficacy | immediately (5 minutes) before and after intervention (relaxation or neurocognitive test battery)
  Participants are subjected to pain measurement, preceded and followed by the collection of saliva samples to analyze cortisol concentrations. Afterwards participants are randomly (by lottery) allocated to group 1 or 2. Group 1 performs a battery of neurocognitive tests and group 2 receives a relaxation session. Afterwards pain measurement with cortisol analyses is repeated.
  One week later the procedure is repeated, while group 1 receives the relaxation session and group 2 performs the neurocognitive test.

SECONDARY OUTCOMES:
neurocognitive performance | once in the study design, immediately (5 minutes) preceded and followed by the pain measurements
  Participants are subjected to pain measurement, preceded and followed by the collection of saliva samples to analyze cortisol concentrations. Afterwards participants are randomly (by lottery) allocated to group 1 or 2. Group 1 performs a battery of neurocognitive tests and group 2 receives a relaxation session. Afterwards pain measurement with cortisol analyses is repeated.
  One week later the procedure is repeated, while group 1 receives the relaxation session and group 2 performs the neurocognitive test.
cortisol response to pain | immediately (1 minute) before and after pain measurements
  Participants are subjected to pain measurement, preceded and followed by the collection of saliva samples to analyze cortisol concentrations. Afterwards participants are randomly (by lottery) allocated to group 1 or 2. Group 1 performs a battery of neurocognitive tests and group 2 receives a relaxation session. Afterwards pain measurement with cortisol analyses is repeated.
  One week later the procedure is repeated, while group 1 receives the relaxation session and group 2 performs the neurocognitive test.

CONTACTS AND LOCATIONS:
Locations (1):
- Vrije Universiteit Brussel, Brussels, Brussels Capital, Belgium